CLINICAL TRIAL: NCT06933290
Title: Effect of Flavored, Carbonated Drinks on Salivary Flow, Salivary Composition, and Taste Perceptions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PEP-2423
Record Dates: First submitted 2025-04-01; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Taste Perception; Saliva Production
Keywords: taste; saliva; food pairing; salivary protein; mucin; salivary flow rate
MeSH Terms: conditions — Medullary cystic kidney disease 1 | interventions — Beverages

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Partially blinded. Uncarbonated flavored drinks and water are distinguishable from carbonated flavored drinks and water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Flavored carbonated drink 1 (Experimental): Flavored carbonated beverage with nutritive sweeteners
  Interventions: Other: Beverage
- Flavored carbonated drink 2 (Experimental): Flavored carbonated beverage with non-nutritive sweeteners
  Interventions: Other: Beverage
- Flavored drink (Experimental): Flavored non-carbonated beverage with nutritive sweeteners
  Interventions: Other: Beverage
- Flavored non-carbonated drink (Experimental): Flavored non-carbonated beverage with non-nutritive sweeteners
  Interventions: Other: Beverage
- Carbonated Water (Experimental): Unflavored carbonated water
  Interventions: Other: Beverage
- Water (Experimental): Plain, unflavored, non-carbonated water
  Interventions: Other: Beverage

INTERVENTIONS:
Other: Beverage — 15 milliliter aliquot interspersed with tastants with a 3 minute break between tastants

SUMMARY:
To determine the effect of flavored, carbonated drinks on salivary flow rate, saliva composition, and taste perceptions compared with control drinks (water, carbonated water, non-carbonated)

DETAILED DESCRIPTION:
Previous studies have shown that drinking a beverage can stimulate the production of saliva and alter its composition. These effects could impact oral processing and taste perceptions. Various ingredients in beverages such as carbonation may affect saliva and oral processing. The objective of this study is to determine the effect of flavored carbonated beverages on salivary flow rate, saliva composition (pH, mucins, carbonic anhydrase, and total protein), and taste perceptions compared with unflavored and non-carbonated control drinks.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female
* If female, subject is not pregnant or nursing (based on self-report)
* Subject is 18-45 years of age, inclusive
* Subject is a regular consumer of carbonated drinks (questionnaire)
* Subject is willing to avoid alcohol consumption 24 hours prior to visits
* Subject is willing to fast (no food or gum) for 2 hours prior to study sessions
* Able to speak, write, and read English
* Provision of written consent to participate

Exclusion Criteria:

* Subject smokes, vapes, or uses any nicotine/tobacco products (or has quit for less than 6 months)
* Subject currently has or recently had an illness (cold, flu, COVID) within the past month
* Subject has a condition affecting the oral cavity such as Xerostomia (dry mouth), Sores/lesions, Untreated dental caries, Major dental implants/appliances (including dentures)
* Subject has a reduced sense of taste (dysgeusia) or smell (parosmia)
* Subject has a health condition that would interfere with the study as indicated on the general health questionnaire (GHQ) (including cardiovascular, renal, or metabolic diseases)
* Subject has participated in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any PepsiCo product. If subject is unsure if a company would be considered a competitor to PepsiCo, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
Salivary flow rate | At each of six 2 hour test sessions 2-8 days apart at same time of day
  5 minute passive drool saliva and 10 minute filter paper saliva (one sample each from tongue and palate) collected in a fixed sequence of tastant flavors (same for each session) and the assigned test beverage intervention (different for each session)

SECONDARY OUTCOMES:
Salivary pH | Sequence of repeated sampling over 2 hours on each of 6 test days with a different beverage and the same tastants each test day
  Lab test
Saliva carbonic anhydrase concentration | Sequence of repeated sampling over 2 hours on each of 6 test days with a different beverage and the same tastants each test day
  Lab test, unit mg/L
Saliva total protein concentration | Sequence of repeated sampling over 2 hours on each of 6 test days with a different beverage and the same tastants each test day
  Lab test, unit mg/ml
Saliva mucin 5B concentration Saliva mucin 5B concentration | Sequence of repeated sampling over 2 hours on each of 6 test days with a different beverage and the same tastants each test day
  Lab test, unit micrograms/ml
Saliva mucin 7 concentration | Sequence of repeated sampling over 2 hours on each of 6 test days with a different beverage and the same tastants each test day
  Lab test, unit micrograms/ml
Taste perceptions | Sequence of repeated sampling over 2 hours on each of 6 test days with a different beverage and the same tastants each test day.
  Labeled Magnitude Scale (LMS)) of intensity of perception rated from barely detectable to strongest imaginable (tastants such as sweet, sour, salty, bitter, umami).
Beverage liking | Sequence of repeated sampling over 2 hours on each of 6 test days with a different beverage and the same tastants each test day
  9-point hedonic scale rating from 1=Dislike extremely to 9= Like extremely
Adverse Events | Symptoms reported at each test day and between visits from Screening to test day six
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, PhD, Principal Investigator — PepsiCo, Inc. Sports Science
Locations (1):
- Gatorade Sports Science Institute, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: No